CLINICAL TRIAL: NCT06830681
Title: A Growth, Tolerability, and Safety Study of a Novel Extensively Hydrolyzed Formula (eHF) in Infants With Cow's Milk Protein Allergy (CMPA)
Brief Title: CMPA-GO Study: Growth and Safety Outcomes in Infants With CMPA Fed a Novel Extensively Hydrolyzed Formula
Acronym: CMPA-GO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision/strategic reason
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2317.CLI
Record Dates: First submitted 2025-01-15; First posted 2025-02-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cow Milk Protein Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formula (Experimental): New generation eHF
  Interventions: Dietary Supplement: New generation eHF
- Control Formula (Active Comparator): Commercial eHF
  Interventions: Dietary Supplement: Commercial eHF

INTERVENTIONS:
Dietary Supplement: New generation eHF — New generation of a whey-based eHF formula intended for the dietary management of infants with CMPA.
  Arms: Test Formula
Dietary Supplement: Commercial eHF — Commercial whey-based eHF formula intended for the dietary management of infants with CMPA.
  Arms: Control Formula

SUMMARY:
CMPA-GO Study: Growth and safety Outcomes in infants with CMPA fed a novel extensively hydrolyzed formula

ELIGIBILITY:
Inclusion Criteria:

1. Full term infant (gestational age ≥37 weeks and ≤42 weeks).
2. Birth weight ≥2500 g and ≤4500 g.
3. Infant aged ≥29 days (>4 weeks) and <5 months (≤22 weeks).
4. Not breastfed at time of Screening Visit.
5. History of an immediate-type (IgE-mediated) allergic reaction to a cow's milk-containing food or at least 2 persistent severe symptoms suggestive of delayed-onset (non-IgE-mediated) CMPA.

Exclusion Criteria:

1. Prior use of eHF, HRF or AAF for more than 2 weeks before randomization.
2. Demonstrated chronic malabsorption not due to CMPA.
3. History of anaphylaxis to CMP.
4. Participants with a history of confirmed Food Protein-induced Enterocolitis Syndrome (FPIES) or Heiner syndrome.
5. Any contraindication to the open OFC (eg. unstable respiratory disease), or any disorder in which epinephrine is contraindicated.
6. History of any immunotherapy for CMPA.
7. Past or current disease or disorder which, in the opinion of the Investigator or the sponsor either places the participant at risk because of participating in the study or may influence the results of the study, or the subject's ability to participate in the study.

Ages: 4 Weeks to 22 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Growth | 16 weeks
  To assess the growth by body weight (in g), body length (in cm) and head circumference (in cm) of infants fed with the Test formula, compared to infants fed with the Control formula over 16 weeks of formula use.

SECONDARY OUTCOMES:
Safety via reporting of adverse events (AEs) and serious adverse events (SAEs) | 52 weeks
  Data gathered by monitoring adverse events with relatedness, seriousness, and severity over 52 weeks.
Tolerability | 52 weeks
  Tolerability of the formulas assessed by the Infant Gastrointestinal Symptom Questionnaire (IGSQ) and and Cow's Milk-related Symptom Score (CoMiSS®).
Growth | 52 weeks
  The growth by body weight (in g), body length (in cm) and head circumference (in cm) of infants over 52 weeks.
Stool frequency and characteristics | 52 weeks
  Stool frequency and characteristics over 52 weeks based on Brussels Infant and Toddler Stool Scale (BITSS).
Quality of life | 52 weeks
  Quality of life over 52-weeks assessed by by 2 validated QoL scales ("Infant and Toddler Quality of Life" [ITQOL] and 'Food hypersensitivity famiLy ImPact' [FLIP]).

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Pediátrico Uncibay, Málaga, Spain